CLINICAL TRIAL: NCT07310316
Title: A Retrospective Cohort Study : Efficacy and Safety of Variceal Embolization Combined With Partial Splenic Artery Embolization in the Treatment of Variceal Bleeding in Cavernous Transformation of Portal Vein.
Brief Title: Efficacy and Safety of Variceal Embolization Combined With Partial Splenic Artery Embolization for Variceal Bleeding in Cavernous Transformation of Portal Vein.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Tie Jun, Director of clinical research, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252459-F-1
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cavernous Transformation of Portal Vein; Gastroesophageal Varices Bleeding
Keywords: Cavernous Transformation of Portal Vein; Esophageal and gastric variceal bleeding; Variceal Embolization; Partial Splenic Artery Embolization
MeSH Terms: conditions — Portal Vein, Cavernous Transformation Of

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTPV (Experimental): A minority of CTPV patients with well-established collateral circulation may remain asymptomatic. However, the majority develop complications of portal hypertension, such as esophagogastric variceal bleeding, ascites, and hypersplenism. Variceal bleeding in particular is characterized by acute onset and high mortality.
  Interventions: Procedure: Variceal Embolization Combined With Partial Splenic Artery Embolization

INTERVENTIONS:
Procedure: Variceal Embolization Combined With Partial Splenic Artery Embolization — Variceal Embolization :
  1. Under ultrasound guidance, a branch of the portal or splenic vein was percutaneously punctured.
  2. Angiography was performed with pressure measurements to evaluate the varices.
  3. The varices were embolized using spring coils and/or tissue adhesive .
  4. Post-embolization angiography was subsequently performed to assess the technical outcome.
  Partial Splenic Artery Embolization :
  1. The right femoral artery was punctured using the Seldinger technique.
  2. Digital subtraction angiography (DSA) was performed following selective catheterization of the splenic artery to delineate its anatomy and branching pattern.
  3. Embolic particles were injected under fluoroscopic guidance.
  4. Intermittent follow-up splenic arteriography was performed, on the basis of the reduction in blood flow velocity, to evaluate the degree of embolization.
  5. The range of the embolization was targeted at 50-60% of the splenic parenchyma.

SUMMARY:
The management of variceal bleeding in patients with cavernous transformation of portal vein (CTPV) generally adheres to the principles applied to cirrhotic portal hypertension, including pharmacological therapy, endoscopic intervention, transjugular intrahepatic portosystemic shunt (TIPS), and surgery. However, the distinct hemodynamic profile caused by portal vein occlusion in CTPV introduces specific therapeutic challenges: 1. Conventional pharmacological and endoscopic treatments often yield suboptimal outcomes. 2. Splenectomy with periesophagogastric devascularization is associated with significant complication rates and elevated perioperative mortality. 3. The feasibility of TIPS depends on sufficient portal venous inflow to ensure stent patency, while also carrying a risk of hepatic encephalopathy. Based on these considerations, the investigators hypothesize that for patients with extensive portal thrombosis and inadequate portal inflow who are ineligible for TIPS, a combination of variceal embolization and partial splenic artery embolization may reduce portal pressure and decrease the risk of esophagogastric variceal bleeding. To evaluate this hypothesis, a retrospective cohort study has been designed.

DETAILED DESCRIPTION:
Cavernous transformation of the portal vein (CTPV) is primarily caused by portal vein thrombosis (PVT). It is characterized by the formation of a network of tortuous, dilated, and malformed venous channels around the obstructed portal vein-a morphology that macroscopically resembles a sponge, hence the name. While a minority of patients with well-developed collateral circulation may remain asymptomatic, most develop complications of portal hypertension, such as esophagogastric variceal bleeding, ascites, and hypersplenism. Variceal bleeding, in particular, is associated with acute onset and high mortality. The management of variceal bleeding in CTPV generally follows guidelines for cirrhotic portal hypertension, including pharmacological therapy, endoscopic treatment, transjugular intrahepatic portosystemic shunt (TIPS), and surgical intervention. However, the distinct hemodynamics resulting from portal vein occlusion pose specific therapeutic challenges:

1. Limited Efficacy of Conventional Pharmacological and Endoscopic Therapies: The chronic organic obstruction in CTPV renders pharmacological agents that reduce portal pressure-such as non-selective beta-blockers-largely ineffective, as they cannot adequately decrease pressure distal to the occlusion. Furthermore, the extensive and complex collateral circulation that develops (e.g., gastroesophageal varices, retroperitoneal venous networks) is often multifocal and highly interconnected. This makes it difficult for endoscopic band ligation or sclerotherapy to comprehensively address all potential bleeding sources. As a result, CTPV patients experience significantly higher rebleeding rates after endoscopic therapy compared to those with conventional portal hypertension.
2. Challenges of Splenectomy with Periesophagogastric Devascularization: Although this classic surgical procedure is used for variceal bleeding in standard portal hypertension, its application in CTPV is complicated by several factors. The spleen is often markedly enlarged and adherent to adjacent structures due to chronic congestion, and the splenic hilar vessels are tortuous and friable, increasing the risk of intraoperative hemorrhage. Moreover, the abundant collateral circulation requires the ligation of a much larger number of vessels than in typical cases. Incomplete devascularization can lead to rebleeding, while the extensive nature of the surgery-coupled with chronic malnutrition and reduced hepatic reserve-elevates the risks of infection, liver failure, and thrombosis, contributing to high perioperative mortality.
3. Limitations of TIPS: While TIPS has shown efficacy in selected CTPV patients with portal hypertension, its success depends on sufficient portal venous inflow to maintain stent patency. In cases with extensive thrombosis involving the splenic or superior mesenteric veins, inadequate inflow increases the risk of early stent thrombosis and shunt dysfunction. Additionally, TIPS carries a well-established risk of hepatic encephalopathy, necessitating careful patient selection, particularly in those with advanced liver dysfunction (Child-Pugh class C) or high baseline encephalopathy risk.

Evidence suggests that combined variceal embolization and partial splenic artery embolization achieves hemostatic outcomes comparable to modified TIPS in cirrhotic portal hypertension, with similar rebleeding rates. This dual interventional approach may also confer benefits in terms of liver function improvement and could be particularly advantageous for patients at high risk of hepatic encephalopathy or with significant liver impairment. Therefore, the investigators hypothesize that for CTPV patients with extensive portosystemic thrombosis and insufficient portal inflow who are unsuitable for shunt procedures, this combined embolization therapy may reduce portal pressure and mitigate the risk of esophagogastric variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. Diagnosis of cavernous transformation of the portal vein (CTPV) confirmed by at least one imaging modality (ultrasonography, CT, or MRI);
3. Portal vein thrombosis (PVT) extending to the splenic vein (SV) and superior mesenteric vein (SMV);
4. History of portal hypertension complicated by variceal bleeding, with recurrent bleeding despite pharmacological and endoscopic therapies;
5. Treated with combined variceal embolization and partial splenic artery embolization;
6. Availability of at least one postoperative follow-up examination with documented clinical data and survival status.

Exclusion Criteria:

1. Concomitant malignant tumor;
2. Active infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of gastroesophageal variceal rebleeding. | 12 months
  Clinically significant rebleeding is defined in accordance with the Baveno V consensus criteria and is identified by recurrence of melena or hematemesis accompanied by any of the following: a) requirement for hospitalization; b) need for blood transfusion; c) hemoglobin decrease of ≥3 g/dL; or d) death within 6 weeks.

SECONDARY OUTCOMES:
All-cause rebleeding | 12 months
New or worsening ascites | 12 months
  Defined as an increase of at least one grade in ascites severity on ultrasound (grading criteria: Grade 0 = none, Grade 1 = mild, Grade 2 = moderate, Grade 3 = large), or persistent ascites requiring paracentesis.
Incidence of overt hepatic encephalopathy | 12 months
  Hepatic encephalopathy is classified according to the 2022 European Association for the Study of the Liver (EASL) Clinical Practice Guidelines using the West-Haven criteria. Overt hepatic encephalopathy is defined as grade II or higher.
Liver function | 12 months
  Liver function will be evaluated using the Child-Pugh score (based on bilirubin, albumin, INR, ascites, and hepatic encephalopathy) and the Model for End-Stage Liver Disease (MELD) score. Child-Pugh Score A to C ( scores ranging from 5 to 15), with higher scores indicating more severe liver dysfunction and a worse prognosis. Child-Pugh Score Grading : Class A: 5-6 scores；Class B: 7-9 scores；Class C: 10-15 scores. MELD = 3.78 × Ln[serum total bilirubin (mg/dL)] + 11.2 × Ln[INR] + 9.57 × Ln[serum creatinine (mg/dL)] + 6.4 × (etiology: 0 for cholestatic or alcoholic, 1 for other). Risk Stratification : High Risk: >18 scores; Intermediate Risk: 15-18 scores; Low Risk: ≤14 scores.
Liver transplantation-free survival | 12 months
  Defined as the time from the TIPS procedure to the end of follow-up, liver transplantation, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tie, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes